CLINICAL TRIAL: NCT01400906
Title: A Randomized, Double Blind, Placebo-controlled Three-way Crossover Study in Mild Asthmatics to Evaluate the Effect of Smoking Status on the Attenuation by Inhaled Corticosteroids of the Allergen-induced Asthmatic Response.
Brief Title: Inhalation of Corticosteroids in Smoking and Non-smoking Asthmatics.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 114748
Record Dates: First submitted 2011-07-21; First posted 2011-07-25 (Estimated); Results first posted 2013-09-30 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-06

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- 3 periods cross-over study (Placebo Comparator): Each subject will receive each intervention BID during a 7 days period. The treatment periods are separated by 14 days washout. The sequence in which the interventions are administered are at random and double blind.
  Interventions: Drug: 100 micrograms Fluticasone propionate; Drug: 500 micrograms Fluticasone propionate; Drug: lactose powder

INTERVENTIONS:
Drug: 100 micrograms Fluticasone propionate — 100 micrograms micronized drug blended with lactose in dry powder inhalator
  Other Names: Flixotide
Drug: 500 micrograms Fluticasone propionate — 500 micrograms micronized drug blended with lactose in dry powder inhalator
  Other Names: Flixotide
Drug: lactose powder — lactose powder in dry powder device : placebo comparator

SUMMARY:
People with asthma suffer from breathlessness because the small tubes (bronchioles) that carry air in and out of the lungs become inflamed and narrow. Steroids reduce the inflammation, and are commonly used to control asthma, but they do not work well in some asthmatics, particularly those who smoke.

This study is done to find out more about why smokers with asthma do not benefit from steroid treatment. In this study, the effect of Flixotide (fluticasone propionate), a steroid widely used to treat asthma, is tested in smokers and non-smokers with mild asthma.

16 smokers and 16 non-smokers, aged 18-55 years will be enrolled in this study.

Subjects will take each of the following treatments:

* 100 micrograms Flixotide twice daily for 7 days;
* 500 micrograms Flixotide twice daily for 7 days; and
* placebo (dummy medicine) twice daily for 7 days.

Study design: subjects will have a screening visit (over 2 days), and will take part in 3 treatment periods (which are separated by interval of at least 14 days); a follow-up visit is scheduled 7 days after the last intake of study treatment.

The order in which order the subjects will take the treatments is defined at random. Total study duration: about 11 weeks.

To test the effects of Flixotide, the subject's responses to :

* an inhaled allergen test
* a PC20 methacholine test
* blood, urine and sputum PD markers will be analysed.

This study will take place in 2 centres: 1 in the United Kingdom and 1 in Belgium. The units will recruit participants by advertising (newspaper, radio, and websites), word of mouth, from volunteer databases, and via the centres' websites.

DETAILED DESCRIPTION:
Most patients with asthma are successfully treated with inhaled corticosteroid (ICS) therapy, either alone or in combination with long-acting beta 2-agonists, with minimal or no side effects. However, a significant proportion of asthmatic patients, including present cigarette smokers and former cigarette smokers, fail to respond well to ICS, alone or in combination with other therapies.

In a randomized, placebo-controlled study, the efficacy of inhaled fluticasone propionate (FP), 1000 μg/day on peak expiratory flow (PEF) and bronchial hyper-reactivity in smokers with mild asthma was assessed compared with non-smoking asthmatics. Asthmatics who smoked showed impaired responses to ICS therapy compared with non-smoking asthmatics [Chalmers, 2002] and this lack of responsiveness appears to be dose-dependent. When the dose of ICS is increased, the disparity between lung function, rescue inhaler usage and asthma control seen in smokers and non-smokers decreases [Tomlinson, 2005].

Interestingly, smoking also affects the ability of ICS to suppress exhaled nitric oxide (eNO) levels in asthmatics [Horváth, 2004]. Smoking cessation improves basal lung function but requires at least a year to demonstrate any improvement in Glucocorticoid (GC) responsiveness with respect to morning peak expiratory flow, but not FEV1, after therapy with high-dose oral prednisolone [Chaudhuri , 2006].

Smoking asthmatics have more severe disease requiring more therapy, have more hospital admissions and are more likely to die from asthma [Thomson, 2005].

Cigarette smoking remains therefore one of the commonest causes of steroid resistance in asthma, however many aspects of the development and restoration of corticosteroid resistance remain unclarified in this population partly due to the paucity of studies performed.

The mechanisms underlying GC resistance in smoking asthmatics are incompletely understood but are thought to include noneosinophilic (often neutrophilic) airway inflammation [Chalmers, 2001], impaired corticosteroid receptor function, and/or reduced histone deacetylase activity [Adcock, 2008]. In support of these effects of smoking on asthma, animal models show that smoking can increase inflammation in allergic models of asthma and can affect steroid responsiveness.

Tobacco smoke exposure (4 cigarettes/day for 3weeks) had a small neutrophilic effect in mice, whereas ovalbumin exposure had no inflammatory effect in the airways, but increased allergen-specific IgE [Moerloose, 2006]. More recently in mouse models, cigarette smoke has been shown to enhance T-helper-(TH)2-driven airway inflammation [Van Hove , 2008].

Inhaled allergens are an important trigger of exacerbations in asthma [Johnston, 2006].

The airway inflammation induced by inhaled allergens, and the effects of drugs on this airway inflammation, can be studied using an experimental allergen challenge model. All the currently approved drugs used to treat asthma modify, in some way, allergen-induced airway responses. Following inhalation of the appropriate allergen extract, sensitive subjects, i.e. atopic-asthmatics, develop an acute bronchoconstriction which peaks at 20 to 30 minutes post-allergen and lasts for approximately two hours before recovery.

This early response (EAR) reflects mast cell activation and subsequent release of mainly spasmogenic mediators and correlates with the extent of airway inflammation and disease activity [Grzelewska-Rsymowska, 1995]. In approximately 50% of patients, the EAR is followed by a late-phase asthmatic response (LAR). This more prolonged airway narrowing is associated with influx of activated inflammatory cells, especially eosinophils, into the airways and represents the more chronic features of asthma, consisting of a prolonged airway narrowing through both bronchospasm and airway inflammation.

The sequelae of the LAR can last several days and up to 3 weeks. Also, the late response has been shown to be associated with an increase in airway hyperresponsiveness (AHR) to stimuli, such as methacholine for several days after allergen challenge [Hansel, 2002].

This clinically relevant model of allergic bronchoconstriction has been useful in humans for exploring the time-course of cellular inflammation and the associated physiological changes, particularly related to eosinophils, basophils and dendritic cells [O'Byrne, 2009].In non smoking asthmatics, regular treatment with inhaled corticosteroids has been shown to attenuate the early allergic response, perhaps by reducing the number of mast cells in airways [Gauvreau, 2000] and to improve the late-phase asthmatic response [Kidney, 1997; Cockcroft, 1987].

As previous allergen challenge studies with therapeutic interventions have been conducted only in the population of non-smokers, this study will be the first to examine the allergen challenge response to FP in smoking asthmatics. The primary endpoint of this study will be the degree of attenuation of the late-phase asthmatic response.

ELIGIBILITY:
Inclusion Criteria:

* males and females between 18 and 55 years of age inclusive
* female subject of child-bearing potential and agrees to use one of the contraception methods; or of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum FSH levels > 40 mIU/mL and estradiol < 40 pg/ml (<140 pmol/L) or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy.
* male subjects with female partners of child-bearing potential must agree to use a contraception method
* body weight ≥50 kg and BMI within the range (18.5-35) kg/m2 (inclusive)
* documented history of bronchial asthma, first diagnosed at least 6 months prior to the first screening visit (according to the BTS guideline 2009), and currently being treated only with prn short-acting inhaled β2-agonist therapy
* current smokers or non-smokers or ex-smokers
* pre-bronchodilator FEV1 >70% of predicted at screening
* sensitivity to methacholine with a provocative concentration of methacholine resulting in a 20 % fall in FEV1 of < 8 mg/ml at screening
* able to produce acceptable induced sputum samples
* positive wheal and/or flare reaction (≥ 3 mm relative to negative control) to at least one allergen on skin prick testing at screening or within 12 months of the study start
* screening allergen challenge must demonstrate that the subject experiences both an early and late asthmatic response.
* AST, ALT, alkaline phosphatase and bilirubin <=1.5xULN
* written informed consent
* able to understand and comply with the study procedures, planned treatment period and other protocol requirements and stated restrictions

Exclusion Criteria:

* past or present disease (other than asthma)
* respiratory tract infection and / or exacerbation of asthma within 4 weeks prior the first dose of study drug
* history of life-threatening asthma
* symptomatic with hay fever at screening or predicted to have symptomatic hay fever during the time of the study
* administration of oral or injectable steroids within 5 weeks of the screening visit or intranasal and / or inhaled steroids within 4 weeks of the screening visit
* unable to abstain from other medication, including non-steroidal anti-inflammatory drugs, anti-depressants, anti-histamines, anti-asthma and anti-rhinitis or hay fever medication, other than short acting β2-agonists and paracetamol (up to 4 gram per day) for the treatment of minor ailments (such as headache) from 14 days before screening until the follow-up visit
* unable to abstain from short acting β2-agonists as described in the restriction section of the protocol
* if, after two consecutive administrations of saline, during the allergen challenge at screening, the subject still has a fall of FEV1 of 10%
* a positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result
* clinical significant abnormalities in safety laboratory analysis at screening
* significant abnormality on 12-lead ECG at screening
* the subject is undergoing an allergen desensitisation therapy. Subjects with a positive pre-study drug/alcohol screen
* a history of regular alcohol consumption within 6 months of the screening visit
* a positive test for HIV antibody
* the subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer)
* history of being unable to tolerate or complete methacholine and / or allergen challenge test
* use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication
* unable to abstain from medication or supplements that significantly inhibit the cytochrome P450 subfamily enzyme CYP3A4, including but not limited to antiretrovirals (protease inhibitors - e.g. ritonavir indinavir, nelfinavir, ritonavir, saquinavir); imidazole and triazole anti-fungals (e.g. ketoconazole, itraconazole) and macrolide antibiotics (e.g. clarithromycin, telithromycin) from screening and throughout the study
* consumption of red wine, seville oranges, grapefruit or grapefruit juice from 7 days prior to the first dose of study medication
* history of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that contraindicates their participation
* donation of blood or blood products in excess of 500 mL within a 56 day period
* pregnant females at screening or prior to dosing
* lactating females
* unwillingness or inability to follow the procedures outlined in the protocol
* subject is mentally or legally incapacitated
* urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening (for subjects taking part in the non-smokers group of the study)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-07-20; Primary Completion 2012-12-01 (Actual); Study Completion 2012-12-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Brussels, Belgium
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Adcock IM, Barnes PJ. Molecular mechanisms of corticosteroid resistance. Chest. 2008 Aug;134(2):394-401. doi: 10.1378/chest.08-0440. PMID 18682458
- [Background] Chalmers GW, Macleod KJ, Little SA, Thomson LJ, McSharry CP, Thomson NC. Influence of cigarette smoking on inhaled corticosteroid treatment in mild asthma. Thorax. 2002 Mar;57(3):226-30. doi: 10.1136/thorax.57.3.226. PMID 11867826
- [Background] Chalmers GW, MacLeod KJ, Thomson L, Little SA, McSharry C, Thomson NC. Smoking and airway inflammation in patients with mild asthma. Chest. 2001 Dec;120(6):1917-22. doi: 10.1378/chest.120.6.1917. PMID 11742922
- [Background] Chaudhuri R, Livingston E, McMahon AD, Lafferty J, Fraser I, Spears M, McSharry CP, Thomson NC. Effects of smoking cessation on lung function and airway inflammation in smokers with asthma. Am J Respir Crit Care Med. 2006 Jul 15;174(2):127-33. doi: 10.1164/rccm.200510-1589OC. Epub 2006 Apr 27. PMID 16645173
- [Background] Cockcroft DW, Murdock KY. Comparative effects of inhaled salbutamol, sodium cromoglycate, and beclomethasone dipropionate on allergen-induced early asthmatic responses, late asthmatic responses, and increased bronchial responsiveness to histamine. J Allergy Clin Immunol. 1987 May;79(5):734-40. doi: 10.1016/0091-6749(87)90204-1. PMID 3106449
- [Background] Gauvreau GM, Wood LJ, Sehmi R, Watson RM, Dorman SC, Schleimer RP, Denburg JA, O'Byrne PM. The effects of inhaled budesonide on circulating eosinophil progenitors and their expression of cytokines after allergen challenge in subjects with atopic asthma. Am J Respir Crit Care Med. 2000 Dec;162(6):2139-44. doi: 10.1164/ajrccm.162.6.2001120. PMID 11112128
- [Background] GlaxoSmithKline Document Number GM2003/00619/00 Study ID EL110002. A single-centre, randomised, double-blind, double-dummy, placebo-controlled, 3-period crossover study to evaluate the effect of pre-treatment with repeat doses of GW842470X (6mg inhaled once daily via the Cyclohaler for 7 days) on the allergen induced late asthmatic response in subjects with mild to moderate asthma, using fluticasone propionate (250 mcg twice daily for 7 days) as a positive control. Report Date 24-Jun-2004.
- [Background] GlaxoSmithKline Document Number YM2009/00265/00 Study ID LPA111834. A randomised, double-blind, placebo-controlled, 2-period crossover study to evaluate the effect of treatment with GSK2190915 on the allergen-induced asthmatic response in subjects with mild asthma. Report Date 26-Mar-2010.
- [Background] GlaxoSmithKline Document Number YM2010/00033/00 Study ID SIG110762. A randomised, placebo-controlled, incomplete block, three-way crossover study to evaluate the effect of treatment with repeat inhaled doses of GW870086 on the allergen-induced early and late asthmatic response in subjects with mild asthma. Report Date 10-May-2010.
- [Background] Grzelewska-Rzymowska I, Gondorowicz K, Cieslewicz G, Rozniecki J. [Course of non-specific bronchial reactivity to histamine after bronchospasm induced by allergen challenge in patients with bronchial asthma]. Pneumonol Alergol Pol. 1995;63(5-6):273-80. Polish. PMID 7581057
- [Background] Hansel TT, Erin EM, Barnes PJ. The allergen challenge. Clin Exp Allergy. 2002 Feb;32(2):162-7. doi: 10.1046/j.1365-2222.2002.01309.x. No abstract available. PMID 11929474
- [Background] Horvath I, Donnelly LE, Kiss A, Balint B, Kharitonov SA, Barnes PJ. Exhaled nitric oxide and hydrogen peroxide concentrations in asthmatic smokers. Respiration. 2004 Sep-Oct;71(5):463-8. doi: 10.1159/000080630. PMID 15467323
- [Background] Ito K, Chung KF, Adcock IM. Update on glucocorticoid action and resistance. J Allergy Clin Immunol. 2006 Mar;117(3):522-43. doi: 10.1016/j.jaci.2006.01.032. PMID 16522450
- [Background] Johnston NW, Sears MR. Asthma exacerbations . 1: epidemiology. Thorax. 2006 Aug;61(8):722-8. doi: 10.1136/thx.2005.045161. PMID 16877691
- [Background] Kidney JC, Boulet LP, Hargreave FE, Deschesnes F, Swystun VA, O'Byrne PM, Choudry N, Morris MM, Jennings B, Andersson N, Andreasson A, Cockcroft DW. Evaluation of single-dose inhaled corticosteroid activity with an allergen challenge model. J Allergy Clin Immunol. 1997 Jul;100(1):65-70. doi: 10.1016/s0091-6749(97)70196-9. PMID 9257789
- [Background] Moerloose KB, Robays LJ, Maes T, Brusselle GG, Tournoy KG, Joos GF. Cigarette smoke exposure facilitates allergic sensitization in mice. Respir Res. 2006 Mar 29;7(1):49. doi: 10.1186/1465-9921-7-49. PMID 16571114
- [Background] O'Shaughnessy KM, Wellings R, Gillies B, Fuller RW. Differential effects of fluticasone propionate on allergen-evoked bronchoconstriction and increased urinary leukotriene E4 excretion. Am Rev Respir Dis. 1993 Jun;147(6 Pt 1):1472-6. doi: 10.1164/ajrccm/147.6_Pt_1.1472. PMID 8389108
- [Background] O'Byrne PM, Gauvreau GM, Brannan JD. Provoked models of asthma: what have we learnt? Clin Exp Allergy. 2009 Feb;39(2):181-92. doi: 10.1111/j.1365-2222.2008.03172.x. PMID 19187330
- [Background] Singh D, Petavy F, Macdonald AJ, Lazaar AL, O'Connor BJ. The inhaled phosphodiesterase 4 inhibitor GSK256066 reduces allergen challenge responses in asthma. Respir Res. 2010 Mar 1;11(1):26. doi: 10.1186/1465-9921-11-26. PMID 20193079
- [Background] Thomson NC, Spears M. The influence of smoking on the treatment response in patients with asthma. Curr Opin Allergy Clin Immunol. 2005 Feb;5(1):57-63. doi: 10.1097/00130832-200502000-00011. PMID 15643345
- [Background] Tomlinson JE, McMahon AD, Chaudhuri R, Thompson JM, Wood SF, Thomson NC. Efficacy of low and high dose inhaled corticosteroid in smokers versus non-smokers with mild asthma. Thorax. 2005 Apr;60(4):282-7. doi: 10.1136/thx.2004.033688. PMID 15790982
- [Background] Van Hove CL, Moerloose K, Maes T, Joos GF, Tournoy KG. Cigarette smoke enhances Th-2 driven airway inflammation and delays inhalational tolerance. Respir Res. 2008 May 20;9(1):42. doi: 10.1186/1465-9921-9-42. PMID 18489797
- [Derived] Cahn A, Boyce M, Mistry S, Musani N, Rambaran C, Storey J, Ventresca P, Michel O. Randomized trial of allergen-induced asthmatic response in smokers and non-smokers: effects of inhaled corticosteroids. Clin Exp Allergy. 2015 Oct;45(10):1531-41. doi: 10.1111/cea.12610. PMID 26251958
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 114748 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 114748 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 114748 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114748 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114748 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114748 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114748 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 36 participants were enrolled; however, 1 participant was categorized as a screen failure following randomization and wasn't dosed with study drug. Thus, 35 of the 36 participants enrolled received treatment.
Groups:
- Sequence 1: Placebo, FP 100 µg, FP 500 µg: Participants received placebo, Fluticasone Propionate (FP) 100 micrograms (µg), and FP 500 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments, one inhalation in the morning and evening from Day 1 to 6 and one inhalation in the morning on Day 7, from the Dry Powder Inhaler (DPI). The three treatment periods were separated by a washout period of 14 days.
- Sequence 2: Placebo, FP 500 µg, FP 100 µg: Participants received Placebo, FP 500 µg, and FP 100 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments, one inhalation in the morning and evening from Day 1 to 6 and one inhalation in the morning on Day 7, from the DPI. The three treatment periods were separated by a washout period of 14 days.
- Sequence 3: FP 100 µg, Placebo, FP 500 µg: Participants received FP 100 µg, Placebo, and FP 500 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments, one inhalation in the morning and evening from Day 1 to 6 and one inhalation in the morning on Day 7, from the DPI. The three treatment periods were separated by a washout period of 14 days.
- Sequence 4: FP 100 µg, FP 500 µg, Placebo: Participants received FP 100 µg, FP 500 µg, and Placebo in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments, one inhalation in the morning and evening from Day 1 to 6 and one inhalation in the morning on Day 7, from the DPI. The three treatment periods were separated by a washout period of 14 days.
- Sequence 5: FP 500 µg, Placebo, FP 100 µg: Participants received FP 500 µg, Placebo, and FP 100 µg in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments, one inhalation in the morning and evening from Day 1 to 6 and one inhalation in the morning on Day 7, from the DPI. The three treatment periods were separated by a washout period of 14 days.
- Sequence 6: FP 500 µg, FP 100 µg, Placebo: Participants received FP 500 µg, FP 100 µg, and Placebo in Treatment Periods 1, 2, and 3, respectively. Participants received all treatments, one inhalation in the morning and evening from Day 1 to 6 and one inhalation in the morning on Day 7, from the DPI. The three treatment periods were separated by a washout period of 14 days.
Period: Treatment Period 1
Arm/Group | Sequence 1: Placebo, FP 100 µg, FP 500 µg | Sequence 2: Placebo, FP 500 µg, FP 100 µg | Sequence 3: FP 100 µg, Placebo, FP 500 µg | Sequence 4: FP 100 µg, FP 500 µg, Placebo | Sequence 5: FP 500 µg, Placebo, FP 100 µg | Sequence 6: FP 500 µg, FP 100 µg, Placebo
Started | 6 | 6 | 6 | 6 | 6 | 5
Completed | 6 | 6 | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Sequence 1: Placebo, FP 100 µg, FP 500 µg | Sequence 2: Placebo, FP 500 µg, FP 100 µg | Sequence 3: FP 100 µg, Placebo, FP 500 µg | Sequence 4: FP 100 µg, FP 500 µg, Placebo | Sequence 5: FP 500 µg, Placebo, FP 100 µg | Sequence 6: FP 500 µg, FP 100 µg, Placebo
Started | 6 | 6 | 6 | 6 | 6 | 5
Completed | 6 | 6 | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Sequence 1: Placebo, FP 100 µg, FP 500 µg | Sequence 2: Placebo, FP 500 µg, FP 100 µg | Sequence 3: FP 100 µg, Placebo, FP 500 µg | Sequence 4: FP 100 µg, FP 500 µg, Placebo | Sequence 5: FP 500 µg, Placebo, FP 100 µg | Sequence 6: FP 500 µg, FP 100 µg, Placebo
Started | 6 | 6 | 6 | 6 | 6 | 5
Completed | 6 | 6 | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Sequence 1: Placebo, FP 100 µg, FP 500 µg | Sequence 2: Placebo, FP 500 µg, FP 100 µg | Sequence 3: FP 100 µg, Placebo, FP 500 µg | Sequence 4: FP 100 µg, FP 500 µg, Placebo | Sequence 5: FP 500 µg, Placebo, FP 100 µg | Sequence 6: FP 500 µg, FP 100 µg, Placebo
Started | 6 | 6 | 6 | 6 | 6 | 5
Completed | 6 | 6 | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Sequence 1: Placebo, FP 100 µg, FP 500 µg | Sequence 2: Placebo, FP 500 µg, FP 100 µg | Sequence 3: FP 100 µg, Placebo, FP 500 µg | Sequence 4: FP 100 µg, FP 500 µg, Placebo | Sequence 5: FP 500 µg, Placebo, FP 100 µg | Sequence 6: FP 500 µg, FP 100 µg, Placebo
Started | 6 | 6 | 6 | 6 | 6 | 5
Completed | 6 | 6 | 6 | 6 | 6 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo, FP 100 µg, and FP 500 µg in 1 of 6 Sequences: All participants received one of the following three treatments in one of three treatment periods, one inhalation in the morning and evening from Day 1 to 6 and one inhalation on the morning on Day 7, from the Dry Powder Inhaler (DPI): Placebo; Fluticasone propionate (FP) 100 micrograms (µg); and FP 500 µg. Participants were randomized to receive treatment in one of the six following sequences: (1) Placebo, FP 100 µg, FP 500 µg; (2) Placebo, FP 500 µg, FP 100 µg; (3) FP 100 µg, Placebo, FP 500 µg; (4) FP 100 µg, FP 500 µg, Placebo; (5) FP 500 µg, Placebo, FP 100 µg; (6) FP 500 µg, FP 100 µg, Placebo. The three treatment periods were separated by a washout period of 14 days.
Arm/Group | Placebo, FP 100 µg, and FP 500 µg in 1 of 6 Sequences
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.0 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage (HER) | 1
  American Indian or Alaska Native | 0
  Central/South Asian HER | 2
  Japanese/East Asian HER/South East Asian HER | 1
  Native Hawaiian or other Pacific Islander | 0
  White | 31

OUTCOME MEASURES:

1. Primary Outcome: Late Asthmatic Response (LAR) - Smokers: Absolute Change From Saline in Minimum Forced Expiratory Volume in One Second (FEV1) Between 4-10 Hours (Hrs) After Allergen Challenge on Day 6 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to an allergen 1 hr after dosing on Day 6. Minimum FEV1 over 4-10 hours post-allergen challenge is the minimum value of all of the post-saline time points between 4 and 10 hrs post-allergen challenge, inclusive of the 4 hr and 10 hr timepoints (i.e., minimum over 4 hrs, 4.5 hrs, 5 hrs, 5.5 hrs, 6 hrs, 6.5 hrs, 7 hrs, 7.5 hrs, 8 hrs, 8.5 hrs, 9 hrs, 9.5 hrs, and 10 hrs). Absolute change from saline at each time point was calculated as the highest allergen challenge FEV1 value minus the highest saline FEV1 value. Data were adjusted for the following covariates: period, smoking status, treatment, participant-level Baseline, period-level Baseline, and treatment by smoking status interaction.
Time Frame: Day 6 of each treatment period (up to 11 weeks)
Population: Pharmacodynamic (PD) Population: all participants in the All Subjects Population (all participants who received at least one dose of study medication) who had a post-dose FEV1 assessment in the same period. Only those participants who were smokers were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- Placebo: Participants received placebo, one inhalation in the morning and one in the evening from Day 1 to 6, and one inhalation in the morning on Day 7 from the DPI during one of the three treatment periods. Each treatment period was followed by a washout period of 14 days.
- FP 100 µg: Participants received FP 100 µg, one inhalation in the morning and one in the evening from Day 1 to 6, and one inhalation in the morning on Day 7 from the DPI during one of the three treatment periods. Each treatment period was followed by a washout period of 14 days.
- FP 500 µg: Participants received FP 500 µg, one inhalation in the morning and one in the evening from Day 1 to 6, and one inhalation in the morning on Day 7 from the DPI during one of the three treatment periods. Each treatment period was followed by a washout period of 14 days.
Arm/Group | Placebo | FP 100 µg | FP 500 µg
Number analyzed (Participants) | 16 | 17 | 17
Liters | -0.592 [-0.793 to -0.391] | -0.420 [-0.617 to -0.224] | -0.431 [-0.627 to -0.234]
Statistical Analysis 1: Comparison: Placebo vs FP 100 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.172, 95% CI 2-sided [-0.037 to 0.380] — The estimated value is an adjusted mean difference. Data were adjusted for the following covariates: period, smoking status, treatment, participant-level Baseline, period-level Baseline, and treatment by smoking status interaction
Statistical Analysis 2: Comparison: Placebo vs FP 500 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.161, 95% CI 2-sided [-0.047 to 0.370] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Early Asthmatic Response (EAR): Absolute Change From Saline in Minimum FEV1 and WM FEV1 Between 0-2 Hours (Hrs) After Allergen Challenge on Day 6 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to an allergen 1 hr after dosing on Day 6. Minimum FEV1 over 0-2 hrs post-allergen challenge (Minimum EAR) is the minimum value of all of the post-allergen challenge timepoints up to and including 2 hours post-allergen challenge (i.e., minimum over 5 minutes [min], 10 min, 15 min, 20 min, 30 min, 45 min and 1 hr, 1.5 hrs, and 2 hrs). The WM FEV1 was derived by calculating the area under the curve, and then dividing the value by the relevant time interval. Absolute change from saline at each time point was calculated as the highest allergen challenge FEV1 value minus the highest saline FEV1 value. Data were adjusted for the following covariates: period, smoking status, treatment, participant-level Baseline, period-level Baseline, and treatment by smoking status interaction.
Time Frame: Day 6 of each treatment period (up to 11 weeks)
Population: PD Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the PD Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | FP 100 µg | FP 500 µg
Number analyzed (Participants) | 35 | 35 | 35
Liters
  Minimum FEV1, Smokers, n=16, 17, 17 | -0.799 [-1.020 to -0.579] | -0.769 [-0.986 to -0.551] | -0.817 [-1.034 to -0.600]
  Minimum FEV1, Non-smokers, n=18, 18, 18 | -0.984 [-1.194 to -0.773] | -0.743 [-0.953 to -0.532] | -0.676 [-0.887 to -0.465]
  WM FEV1, Smokers, n=16, 17, 17 | -0.423 [-0.567 to -0.279] | -0.303 [-0.445 to -0.161] | -0.362 [-0.504 to -0.220]
  WM FEV1, Non-smokers, n=18, 18, 18 | -0.531 [-0.669 to -0.394] | -0.349 [-0.486 to -0.211] | -0.311 [-0.448 to -0.173]

3. Secondary Outcome: Absolute Change From Baseline in FEV1 Post-dose on Day 1, Day 6 (Prior to Allergen Challenge), and Day 7
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Baseline FEV1 was measured on Day 1 pre-dose administration. FEV1 was measured on Day 1 post-dose, on Day 6 (prior to allergen challenge), and on Day 7 pre dose administration. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Data were adjusted for the following covariates: period, smoking status, treatment, participant-level Baseline, period-level Baseline, and treatment by smoking status interaction.
Time Frame: Baseline, Day 1, Day 6, and Day 7
Population: PD Population. Only those participants available at the specified time points were analyzed (represented by n=X, X, X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the PD Population.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | FP 100 µg | FP 500 µg
Number analyzed (Participants) | 35 | 35 | 35
Liters
  Day 1, Smokers, n=17, 17, 17 | 0.156 [0.063 to 0.249] | 0.216 [0.123 to 0.309] | 0.177 [0.084 to 0.270]
  Day 6, Smokers, n=16, 17, 17 | -0.081 [-0.166 to 0.003] | 0.016 [-0.067 to 0.098] | 0.032 [-0.050 to 0.115]
  Day 7, Smokers, n=17, 17, 17 | -0.123 [-0.279 to 0.032] | -0.083 [-0.239 to 0.072] | -0.053 [-0.208 to 0.103]
  Day 1, Non-smokers, n=16, 18, 17 | 0.201 [0.107 to 0.294] | 0.237 [0.147 to 0.327] | 0.217 [0.125 to 0.309]
  Day 6, Non-smokers, n=18, 18, 18 | -0.028 [-0.108 to 0.052] | 0.114 [0.034 to 0.194] | 0.058 [-0.022 to 0.138]
  Day 7, Non-smokers, n=18, 18, 18 | -0.341 [-0.492 to -0.190] | -0.079 [-0.230 to 0.072] | 0.012 [-0.138 to 0.163]

4. Secondary Outcome: Provocative Concentration of Methacholine Resulting in a 20% Reduction in FEV1 (PC20) on Day 7 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants inhaled doubling increments of methacholine until a >=20% decrease in FEV1 from the post-saline value was achieved.
Time Frame: Day 7 of each treatment period (up to 11 weeks)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: milligrams per milliliter
Arm/Group | Placebo | FP 100 µg | FP 500 µg
Number analyzed (Participants) | 35 | 35 | 35
milligrams per milliliter
  Smokers, n=16, 17, 17 | 0.579 [0.391 to 0.855] | 1.233 [0.845 to 1.798] | 1.439 [0.985 to 2.100]
  Non smokers, n=18, 17, 18 | 0.514 [0.356 to 0.743] | 1.488 [1.020 to 2.172] | 2.080 [1.441 to 3.001]

5. Secondary Outcome: Concentration of Exhaled Nitric Oxide (eNO) on Day 6 and Day 7 of Each Treatment Period
Description: The concentration of eNO was measured on Day 6 pre-dose and on Day 7 post-study medication administration. eNO was measured 3 times at each time point, and all 3 measurements were recorded. The mean of the 3 measurements was calculated and was used in the derivation of summary statistics.
Time Frame: Day 6 and Day 7 of each treatment period (up to 11 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Parts per billion
Arm/Group | Placebo | FP 100 µg | FP 500 µg
Number analyzed (Participants) | 35 | 35 | 35
Parts per billion
  Day 6, Pre-dose, Smokers, n=16, 17, 17 | 21.117 (15.2894) | 12.718 (6.5018) | 14.049 (14.8450)
  Day 7, Post-dose, Smokers, n=17, 17, 17 | 45.167 (34.8859) | 16.602 (10.5155) | 16.298 (10.8249)
  Day 6, Pre-dose, Non-smokers, n=17, 18, 18 | 62.980 (30.8968) | 37.252 (17.8334) | 32.572 (17.4064)
  Day 7, Post-dose, Non-smokers, n=18, 18, 18 | 98.837 (42.4567) | 42.869 (25.4944) | 34.989 (16.0285)

6. Primary Outcome: LAR - Non-smokers: Absolute Change From Saline in Minimum FEV1 Between 4-10 Hours (Hrs) After Allergen Challenge on Day 6 of Each Treatment Period
Description: as for outcome 1
Time Frame: Day 6 of each treatment period (up to 11 weeks)
Population: PD Population. Only those participants who were non-smokers were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | FP 100 µg | FP 500 µg
Number analyzed (Participants) | 18 | 18 | 18
Liters | -1.034 [-1.225 to -0.843] | -0.396 [-0.587 to -0.205] | -0.373 [-0.563 to -0.182]
Statistical Analysis 1: Comparison: Placebo vs FP 100 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.638, 95% CI 2-sided [0.440 to 0.836] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs FP 500 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.661, 95% CI 2-sided [0.463 to 0.859] — [estimate comment as in outcome 1, analysis 1]

7. Primary Outcome: LAR - Smokers: Absolute Change From Saline in Weighted Mean (WM) FEV1 Between 4-10 Hrs Following Post-treatment Allergen Challenge on Day 6 of Each Treatment Period
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Participants were exposed to an allergen 1 hour after dosing on Day 6. The WM FEV1 was derived by calculating the area under the curve, and then dividing the value by the relevant time interval. LAR WM FEV1 was measured at 4 hrs, 4.5 hrs, 5 hrs, 5.5 hrs, 6 hrs, 6.5 hrs, 7 hrs, 7.5 hrs, 8 hrs, 8.5 hrs, 9 hrs, 9.5 hrs, and 10 hrs post-allergen challenge on Day 6. Absolute change from saline at each time point was calculated as the highest allergen challenge FEV1 value minus the highest saline FEV1 value. Data were adjusted for the following covariates: period, smoking status, treatment, participant-level Baseline, period-level Baseline, and treatment by smoking status interaction.
Time Frame: Day 6 of each treatment period (up to 11 weeks)
Population: PD Population. Only those participants who were smokers were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | FP 100 µg | FP 500 µg
Number analyzed (Participants) | 16 | 17 | 17
Liters | -0.364 [-0.512 to -0.215] | -0.188 [-0.334 to -0.043] | -0.198 [-0.344 to -0.053]
Statistical Analysis 1: Comparison: Placebo vs FP 100 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.175, 95% CI 2-sided [0.018 to 0.333] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs FP 500 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.165, 95% CI 2-sided [0.008 to 0.323] — [estimate comment as in outcome 1, analysis 1]

8. Primary Outcome: LAR - Non-smokers: Absolute Change From Saline in WM FEV1 Between 4-10 Hrs Following Post-treatment Allergen Challenge on Day 6 of Each Treatment Period
Description: as for outcome 7
Time Frame: Day 6 of each treatment period (up to 11 weeks)
Population: PD Population. Only those participants were non-smokers were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | Placebo | FP 100 µg | FP 500 µg
Number analyzed (Participants) | 18 | 18 | 18
Liters | -0.688 [-0.829 to -0.547] | -0.212 [-0.353 to -0.071] | -0.158 [-0.299 to -0.018]
Statistical Analysis 1: Comparison: Placebo vs FP 100 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.476, 95% CI 2-sided [0.326 to 0.627] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs FP 500 µg; Test type: Superiority or Other; Mean Difference (Final Values) = 0.530, 95% CI 2-sided [0.380 to 0.680] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Neutrophil and Eosinophil Cell Counts in Induced Sputum on Day 7 of Each Treatment Period
Description: Sputum induction was performed using hypertonic saline solution to collect an adequate sample of secretions from lungs. The collected sputum was analyzed for neutrophil and eosinophil counts. Sputum induction was performed after methacholine challenge and post-dose administration on Day 7. Zero values are imputed to 0.001 for this analysis. Data were adjusted for the following covariates: period, smoking status, treatment, participant-level Baseline, period-level Baseline, and treatment by smoking status interaction.
Time Frame: Day 7 of each treatment period (up to 11 weeks)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: 10^4 cells per gram of sputum
Arm/Group | Placebo | FP 100 µg | FP 500 µg
Number analyzed (Participants) | 35 | 35 | 35
10^4 cells per gram of sputum
  Eosinophil count, Smokers, n=7, 7, 5 | 0.400 [0.027 to 5.858] | 0.489 [0.030 to 8.020] | 0.459 [0.000 to 444.058]
  Eosinophil count, Non-smokers, n=11, 11, 10 | 6.911 [0.851 to 56.129] | 0.878 [0.105 to 7.356] | 0.144 [0.010 to 2.162]
  Neutrophil count, Smokers, n=7, 7, 5 | 96.231 [44.622 to 207.532] | 50.313 [22.948 to 110.308] | 87.699 [13.432 to 572.592]
  Neutrophil count, Non-smokers, n=11, 11, 10 | 78.768 [43.324 to 143.209] | 49.532 [27.052 to 90.692] | 36.561 [17.389 to 76.869]

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the treatment period (up to 16 weeks).
Description: SAEs and non-serious AEs were reported for members of the All Subjects Population, comprised of all participants who received at least one dose of study medication.
Arm/Group | Placebo | FP 100 µg | FP 500 µg
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 11/35 | 8/35 | 11/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=35) | FP 100 µg (N=35) | FP 500 µg (N=35)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Oral pruritus (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Eye irritation (Eye disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.